CLINICAL TRIAL: NCT02945267
Title: A Randomized, Controlled, Double Blind, Multicenter Study of Nimotuzumab Plus S1 Versus Placebo Plus S1 as Maintenance Treatment in Patients With Advanced or Metastatic Pancreatic Cancer After First-line Treatment
Brief Title: Nimotuzumab Plus S1 Versus Placebo Plus S1 as Maintenance Treatment in Patients With Unresectable Pancreatic Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, yihu, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PC20150423
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Unresectable Pancreatic Cancer
Keywords: Pancreatic Cancer; Unresectable; Maintenance Treatment
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — nimotuzumab; S 1 (combination)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nimotuzumab plus S1 (Experimental): Nimotuzumab Injection:400 mg/w, Intravenous infusion, Infusion time ≥ 60 min, d1, once every two weeks; S1:40 mg (Body surface area<1.5 m2) or 60mg (Body surface area>1.5 m2) ,oral,d1-d14, every three weeks for a cycle
  Interventions: Drug: Nimotuzumab plus S1
- Placebo plus S1 (Active Comparator): Placebo:400 mg/w, Intravenous infusion, Infusion time ≥ 60 min, d1, once every two weeks; S1:40 mg (Body surface area<1.5 m2) or 60 mg (Body surface area>1.5 m2) ,oral,d1-d14, every three weeks for a cycle
  Interventions: Drug: Placebo plus S1

INTERVENTIONS:
Drug: Nimotuzumab plus S1 — Nimotuzumab Injection: 400 mg/w, Intravenous infusion, Infusion time ≥ 60 min, d1, once every two weeks;S1: 40 mg (Body surface area<1.5 m2) or 60 mg (Body surface area>1.5 m2) ,oral,d1-d14, every three weeks for a cycle
  Other Names: Taixinsheng，Tegafur Gimeracil Oteracil Potassium Capsule
  Arms: Nimotuzumab plus S1
Drug: Placebo plus S1 — Placebo: 400 mg/w, Intravenous infusion, Infusion time ≥ 60 min, d1, once every two weeks;S1: 40 mg (Body surface area<1.5 m2) or 60 mg (Body surface area>1.5 m2) ,oral,d1-d14, every three weeks for a cycle
  Other Names: Tegafur Gimeracil Oteracil Potassium Capsule
  Arms: Placebo plus S1

SUMMARY:
Background: Monotherapy with S-1, oral fluoropyrimidine, shows non-inferiority to gemcitabine in overall survival (OS) with good tolerability for advanced pancreatic cancer in Asian patients. It is also shown that nimotuzumab plus gemcitabine could improve OS and progression free survival (PFS) in patients with unresectable pancreatic cancer. However, it is still unknown whether nimotuzumab plus S1 would improve more to OS and PFS than single S-1. Maintenance treatment, as a new treatment pattern, has also been tried in these patients after first line treatment to improve the OS. Thus, this study is designed to compare nimotuzumab plus S1 to placebo plus S1 as maintenance treatment in patients with locally advanced or metastatic pancreatic cancer who has benefited from the first-line treatment of gemcitabine combined with nimotuzumab and S1 (complete response+partial response+stable disease).

Patients and methods: 60 patients will be enrolled,and randomized in a 1:1 ratio to group nimotuzumab plus S1 and group placebo plus S1. nimotuzumab/placebo: 400 mg/w, intravenous infusion, Infusion time ≥ 60 min, d1, once every two weeks. S1: oral, 40 mg (Body surface area<1.5 m2) or 60 mg (Body surface area>1.5 m2), d1-d14, every three weeks for a cycle. Treatment interventions will be stopped under the conditions of disease progression or intolerable toxic reaction or participants ask to quit. The primary endpoint is the time to disease progression since randomization (TTP), secondary points include OS, 3 years overall survival rate (OSR) and safety.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years;
* Karnofsky Performance Status≥ 60;
* histologically proven locally advanced or metastatic pancreatic cancer,and unsuitable for radiotherapy or surgery resection;
* benefited from the first line treatment of gemcitabine plus nimotuzumab and S1 (complete response+partial response+stable disease);
* at least 4 weeks from the end of the first-line treatment;
* with at least 1 measurable and evaluable lesion;
* anticipated over survival≥12 weeks;
* AST/ALT≤2.5 ULN (≤5 ULN for patients with hepatic metastases); total bilirubin≤2 ULN （≤3 ULN for patients with hepatic metastases); neutrophil count≥1.5×109/L; platelet counts≥100×109/L; hemoglobin level≥90 g/L; creatinine clearance rate≥ 60 mL/min
* written informed consent

Exclusion Criteria:

* previously received the following treatments: anticancer chemotherapy/molecularly targeted therapy as palliative treatment, or targeted chemotherapy and no progression, another interventional clinical trail within 4 weeks;
* underwent major surgery within 4 weeks;
* with brain or leptomeningeal metastases;
* history of malignancy other than pancreatic cancer;
* presented symptomatic abdominal fluid and needed treatment;
* with other serious diseases such as diabetes,active infection;
* known for allergy to anti epidermal growth factor receptor antibody

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
TTP | 3 years

SECONDARY OUTCOMES:
OS | 3 years
OSR | 1-3 years
Adverse Events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yi Hu, PhD, Principal Investigator — Chinese PLA General Hospital
Locations (7):
- China (7):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - First Affiliated Hospital of PLA General Hospital, Beijing
  - Rocket Army General Hospital, PLA, Beijing
  - The 306TH Hospital of PLA, Beijing
  - Air Force General Hospital, PLA, Beijing
  - Beijing Hospital, Beijing
  - Chinese PLA General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes